CLINICAL TRIAL: NCT05160961
Title: Comparison of the Effects of Ultrasound-guided Serratus Anterior Plane Block and Erector Spinae Plane Block on Postoperative Acute and Chronic Pain for Patients Who Underwent Video-assisted Thoracoscopic Surgery.
Brief Title: US-Guided SAPB Versus ESPB on Acute and Chronic Pain After VATS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.Kurul-E1-21-2142
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain; Video-Assisted Thoracoscopic Surgery; Serratus Anterior Plane Block; Erector Spinae Plane Block; Acute Pain; Chronic Pain
Keywords: Serratus anterior plane block; Erector spinae plane block; Acute Pain; Chronic Pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Anterior Plane Block (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle will be advanced via the in-plane technique beneath the serratus anterior muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 20 ml 0.25% bupivacaine will be injected into the area.
  Interventions: Procedure: Serratus anterior plane block
- Erector spinae plane block (Active Comparator): After the linear ultrasound (US) probe will be placed 2-3 cm lateral to the T5 spinous process, 20 ml of 0.25% bupivacaine hydrochloride will be injected into the interfacial space below the erector spinae muscle, above the transverse process.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Serratus anterior plane block — Serratus anterior plane block will be performed unilaterally, under US guidance, before the surgical operation, after the induction of anesthesia, when the patient is placed in the lateral decubitus position.
  Other Names: Drug
  Arms: Serratus Anterior Plane Block
Procedure: Erector spinae plane block — Erector spinae plane block will be performed unilaterally, under US guidance, before the surgical operation, after the induction of anesthesia, when the patient is placed in the lateral decubitus position.
  Other Names: Drug
  Arms: Erector spinae plane block

SUMMARY:
Postoperative acute and chronic pain is frequently observed in patients undergoing video assisted thoracoscopic surgery (VATS). This prolongs the discharge time of patients and increases the frequency of postoperative pulmonary complications. Recently, alternative analgesic methods such as thoracic paravertebral block (TPVB), erector spinae plane block (ESPB), and serratus anterior plane block (SAPB) which are thought to have less side effects than thoracic epidural analgesia, have been used. Among these methods, ultrasound (US) guided TPVB is the most preferred method. In addition, ESPB and SAPB application is increasing in patients undergoing VATS. In the literature, the number of cases performed with ESPB and SAPB and randomized controlled prospective studies with ESPB and SAPB are increasing. In this study, it is planned to compare the effects of US-guided SAPB and ESPB on postoperative acute and chronic pain in patients undergoing VATS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* American Society of Anesthesiologists physical status I-II-III
* Body mass index between 18-30 kg/m2
* Patients undergoing elective video assiste thoracoscopic surgery

Exclusion Criteria:

* Advanced cancer
* History of chronic analgesic therapy
* History of local anesthetic allergy
* Infection in the intervention area
* Patients with bleeding disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Pain scores | First 24 hours after surgery
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 1st, 2nd, 4th, 8th, 16th and 24th hours after surgery.

SECONDARY OUTCOMES:
Chronic pain | 3rd month and 6th month
  Chronic pain findings will be evaluated in the 3rd month and 6th month after surgery by using visual analog from 0 (no pain) to 10 (worst pain). Neuropathic pain symptoms (Burning, stabbing, or electric shock-like pain; tingling, numbness, or a "pins and needles" feeling, hyperalgesia, allodynia and hypoesthesia) will also be asked to the participants in the 3rd month and 6th month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Zengin, MD, Principal Investigator — Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No